CLINICAL TRIAL: NCT03575572
Title: Colchicine in Postoperative Fontan Patients (CPFP)
Brief Title: Colchicine in Postoperative Fontan Patients
Acronym: CPFP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Staffing changes impacted by COVID-19 pandemic resulting in inadequate personnel to facilitate study.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Stephanie Goldstein, House Officer, Pediatric Cardiology and House Officer, Pediatric Critical Care (during active trial status), University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00143571
Record Dates: First submitted 2018-06-18; First posted 2018-07-02 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Single-ventricle; Heart Diseases
Keywords: Fontan; Colchicine; heart surgery
MeSH Terms: conditions — Univentricular Heart; Heart Diseases | interventions — Colchicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Colchicine (Experimental): Colchicine will be given at 0.6 mg once daily for the duration of chest tube output plus 24 hours after chest tube removal with a maximum of 4 weeks duration.
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Colchicine is an alkaloid approved in 1961 for the use in Familial Mediterranean Fever in adults and children 4 years of age or older. It has been widely used for decades in other indications, such as Gout, recurrent pericarditis, pericardial effusions and other inflammatory diseases. This drug is commercially available and is approved in children 4 years and older.

SUMMARY:
The investigators found that there is inflammation in the chest drainage in patients after the Fontan operation. The investigators want to test the theory that Colchicine, an anti- inflammatory medication, can decrease the inflammation in the chest tube drainage after the Fontan operation, and can decrease the amount of time that patients having this surgery will have drainage.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20 months to 5 years and 364 days are eligible
* Diagnosed with single ventricle heart disease requiring Fontan palliation
* Undergoing Fontan palliation at the University of Michigan Congenital Heart Center
* Ability to take oral or enteral medication

Exclusion Criteria:

* Treatment with another investigational drug within 3 months
* Pre-existing myelosuppression or decreased bone marrow activity.
* Current or recent treatment with certain drugs
* Renal or hepatic impairment deemed by the study team
* Conditions and/or post-operative complications that would increase risk to the patient such as mechanical support (ECMO) or issues in the intensive care unit (ICU)

Ages: 20 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Goldstein, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldstein SA, Nolan K, Marchetti K, Stoscup JK, Clewis H, Jarvis K, Halligan NLN, Dahmer MK, Schumacher KR, Rocchini A. Colchicine in post-operative Fontan patients. Cardiol Young. 2023 Jun;33(6):910-916. doi: 10.1017/S104795112200186X. Epub 2022 Jun 20. PMID 39625244

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 people who were consented didn't actually begin the trial. Under the protocol, historical controls were not considered enrolled in this study, so they are not included in participant flow. Historical control data were taken from an observational study with no intervention that was published prior to first enrollment in this trial. Data on the historical controls are available at PMID: 30710164.
Groups:
- Colchicine: All patients entered the intended protocol where Colchicine was empirically given 0.6mg once daily to postoperative Fontan patients starting on postoperative day 2 and ending 1 day after chest tubes were removed or for a maximum of 4 weeks.
Period: Overall Study
Arm/Group | Colchicine
Started (Started is defined here to mean first sample collected.) | 9
Completed | 5
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- Historical Controls: Historical Controls were post-operative Fontan patients who underwent their operation at the University of Michigan. They were part of a prospective observational study that was published in 2019 which included the chest tube drainage sample collection similar to that done with the Colchicine cohort in this trial.
- Total: Total of all reporting groups
Arm/Group | Colchicine | Historical Controls | Total
Number analyzed (Participants) | 9 | 25 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.7 [2.1 to 4.3] | 2.5 [2.1 to 2.9] | NA [NA to NA] — Complete historical control age data is no longer available. So, while median (2.5) and Inter-Quartile Range (2.1 to 2.9) is available for historical controls from previously published data, it is not possible to submit the results without the full population median and inter-quartile range computed. The full data set for the historical controls is not available to recompute the medians and IQR for the two populations combined.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 4 | 18 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 22 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 9 | 25 | 34
Primary Diagnosis [Number; unit: participants]
  Hypoplastic left heart syndrome (HLHS) | 6 | 14 | 20
  Not HLHS | 3 | 11 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Cytokine Total Mass in Pleural Fluid From Patients Treated With Colchicine
Description: Cytokine total mass measured by the Bio-rad Bio-Plex ProHuman Cytokine 17-plex Assay.
Time Frame: Postoperative day 1 ; day most distal from surgery, approximately 7 days after surgery
Measure: Median (Inter-Quartile Range); unit: picograms
Groups:
- Colchicine Per Protocol: All patients entered the intended protocol where Colchicine was empirically given 0.6mg once daily to postoperative Fontan patients starting on postoperative day 2 and ending 1 day after chest tubes were removed or for a maximum of 4 weeks.
  These participants completed the protocol.
Arm/Group | Colchicine Per Protocol
Number analyzed (Participants) | 5
picograms
  Interleukin (IL)-8; post op. Day 1 | 60925.8 [27396.7 to 123151.56]
  IL-8, Day 7 | 8684.57 [2346.135 to 19715.275]
  Tumor Necrosis Factor (TNF)-alpha, Day 1 | 6552.7 [4954.770 to 7482.8]
  TNF-alpha, Day 7 | 694.575 [479.288 to 909.863]
  Macrophage Inflammatory Protein (MIP)-1 Beta Day 1 | 4949.89 [4450.56 to 13543.4]
  MIP-1 Beta Day 7 | 247.775 [225.088 to 270.463]
  Interleukin (IL)-10 Day 1 | 5286.55 [4560.4 to 9763.27]
  IL-10 Day 7 | 132.755 [117.558 to 147.953]

2. Primary Outcome: Difference in Change of Cytokine Concentrations in Pleural Fluid Patients Treated With Colchicine Compared to Historical Controls
Description: Difference is shown via two columns of separate data, but given that enrollment didn't meet target before termination statistical analysis was not done for this measure
Time Frame: Postoperative day 1 ; day most distal from surgery, approximately 7 days after surgery
Measure: Median (Inter-Quartile Range); unit: picograms
Groups:
- Colchicine: All patients entered the intended protocol where Colchicine was empirically given 0.6mg once daily to postoperative Fontan patients starting on postoperative day 2 and ending 1 day after chest tubes were removed or for a maximum of 4 weeks.
  These participants completed the protocol.
Arm/Group | Colchicine | Historical Controls
Number analyzed (Participants) | 5 | 25
picograms
  IL-8 Day 1 | 60925.80 [27396.70 to 123151.56] | 83263.45 [42239.05 to 369274.25]
  IL-8 Day 7 | 8684.57 [2346.14 to 19715.28] | 64695.50 [28829.240 to 253569.74]
  TNF-Alpha Day 1 | 6552.70 [4954.77 to 7482.80] | 8080.38 [6269.6 to 11148.0]
  TNF-ALpha Day 7 | 694.575 [479.288 to 909.863] | 3320.97 [1872.72 to 5481.28]
  MIP-1 Beta Day 1 | 4949.89 [4450.56 to 13543.40] | 11527.80 [6800.60 to 18611.90]
  MIP-1Beta Day 7 | 247.775 [225.088 to 270.463] | 5986.4 [3251.41 to 12216.24]
  IL-10, Day 1 | 5286.55 [4560.4 to 9763.27] | 14474.4 [8099.82 to 25592.7]
  IL-10, Day 7 | 132.755 [117.558 to 147.953] | 885.04 [693.12 to 1665.66]

3. Secondary Outcome: Cytokine Total Mass as Measured in Postoperative Fontan Patients Treated Empirically With Colchicine
Description: Particularly Cytokine total mass of TNF-α, MIP-1β, IL-8, and IL-10, determined by the Bio-rad Bio-Plex ProHuman Cytokine 17-plex Assay
  Data was only collected while patients had chest tubes in place (up to 7 days only)
Time Frame: Postoperative days 1, 2, 3, 4, 7
Measure: Median (Inter-Quartile Range); unit: picograms
Arm/Group | Colchicine Per Protocol
Number analyzed (Participants) | 5
picograms
  IL-8 Day 1 | 60925.80 [27396.70 to 123151.56]
  IL 8 Day 2 | 22178.00 [11356.16 to 57721.6]
  IL 8 Day 3 | 26837.20 [15517.8 to 80660.56]
  IL 8 Day 4 | 50895.36 [17402.06 to 113591.7]
  IL 8 Day 7 | 8684.57 [2346.14 to 19715.28]
  IL 10 Day 1 | 5286.55 [4560.40 to 9763.27]
  IL 10 Day 2 | 2788.44 [2194.92 to 3084.90]
  IL 10 Day 3 | 586.50 [401.60 to 1033.60]
  IL 10 Day 4 | 448.06 [318.24 to 593.46]
  IL 10 Day 7 | 132.755 [117.558 to 147.953]
  TNF Alpha Day 1 | 6552.70 [4954.77 to 7482.80]
  TNF Alpha Day 2 | 6220.50 [2854.30 to 6932.60]
  TNF Alpha Day 3 | 3791.84 [2108.68 to 4360.80]
  TNF Alpha Day 4 | 2517.90 [1248.72 to 2950.66]
  TNF Alpha Day 7 | 694.575 [479.288 to 909.863]
  MIP-1 Beta Day 1 | 4949.89 [4450.56 to 13543.40]
  MIP-1 Beta Day 2 | 3066.80 [2566.10 to 10702.90]
  MIP-1 Beta Day 3 | 4031.04 [2107.66 to 6968.00]
  MIP-1 Beta Day 4 | 2730.50 [2327.64 to 5768.16]
  MIP-1 Beta Day 7 | 247.775 [225.088 to 270.463]

4. Secondary Outcome: Difference in Cytokine Total Mass, as Measured in Postoperative Fontan Patients Treated Empirically With Colchicine in Comparison to a Cohort of Postoperative Fontan Patients
Description: Cytokine total mass measured by Bio-rad Bio-Plex ProHuman Cytokine 17-plex Assay
  Data was only collected from Colchicine patients while they had chest tubes in place (up to 7 days). For historical controls data was collected up through Day 10
Time Frame: Postoperative days 1, 2, 3, 4, 7, 10
Population: Day 10 data was not gathered from participants per protocol, but it was available for historical controls.
Measure: Median (Inter-Quartile Range); unit: picograms
Arm/Group | Colchicine Per Protocol | Historical Controls
Number analyzed (Participants) | 5 | 25
picograms
  IL-8 Day 1 | 60925.80 [27396.70 to 123151.56] | 83263.45 [42239.05 to 369274.25]
  IL-8 Day 2 | 22178.00 [11356.16 to 57721.6] | 50734.56 [20064.46 to 177356.64]
  IL-8 Day 3 | 26837.20 [15517.80 to 80660.56] | 36175.15 [14641.888 to 95957.95]
  IL-8 Day 4 | 50895.36 [17402.06 to 113591.7] | 52203.825 [21544.800 to 142966.54]
  IL-8 Day 7 | 8684.57 [2346.14 to 19715.28] | 64695.5 [28829.24 to 253569.74]
  IL-8 Day 10: number analyzed (Participants) | 0 | 25
  IL-8 Day 10 |  | 140165.900 [28829.240 to 253569.740]
  IL-10 Day 1 | 5286.55 [4560.4 to 9763.27] | 14474.4 [8099.82 to 25592.7]
  IL-10 Day 2 | 2788.440 [2194.92 to 3084.90] | 5341.80 [2882.88 to 9084.43]
  IL-10 Day 3 | 586.59 [401.60 to 1033.60] | 1192.29 [914.91 to 3959.96]
  IL-10 Day 4 | 448.06 [318.24 to 593.46] | 1462.22 [645.84 to 2533.72]
  IL-10 Day 7 | 132.755 [117.558 to 147.953] | 885.04 [693.12 to 1665.66]
  IL-10 Day 10: number analyzed (Participants) | 0 | 25
  IL-10 Day 10 |  | 417.80 [397.70 to 879.52]
  TNF Alpha Day 1 | 6552.70 [4954.77 to 7482.80] | 8080.38 [6269.60 to 11148.00]
  TNF Alpha Day 2 | 6220.50 [2854.30 to 6932.60] | 4761.36 [3666.30 to 8852.98]
  TNF Alpha Day 3 | 3791.84 [2108.68 to 4360.80] | 3495.45 [2314.73 to 5610.040]
  TNF Alpha Day 4 | 2517.90 [1248.72 to 2950.66] | 3411.555 [1894.673 to 6369.735]
  TNF Alpha Day 7 | 694.575 [479.288 to 909.863] | 3320.97 [1872.72 to 5481.28]
  TNF Alpha Day 10: number analyzed (Participants) | 0 | 25
  TNF Alpha Day 10 |  | 2361.60 [1741.88 to 3880.690]
  MIP-Beta Day 1 | 4949.89 [4450.56 to 13543.400] | 11527.80 [6800.60 to 18611.90]
  MIP-Beta Day 2 | 3066.80 [2566.10 to 10702.90] | 8822.96 [5286.89 to 14864.72]
  MIP-Beta Day 3 | 4031.04 [2107.66 to 6968.00] | 6594.00 [3215.19 to 8202.60]
  MIP-Beta Day 4 | 2730.50 [2327.64 to 5768.16] | 7375.96 [2856.50 to 13588.94]
  MIP-Beta Day 7 | 247.775 [225.088 to 270.463] | 5986.40 [3251.41 to 12216.24]
  MIP-Beta Day 10: number analyzed (Participants) | 0 | 25
  MIP-Beta Day 10 |  | 8957.13 [4132.15 to 17056.82]

5. Secondary Outcome: Duration of Pleural Drainage as Measured in Postoperative Fontan Patients Treated Empirically With Colchicine
Description: Duration is measured in days, from date of Fontan surgery to chest tube drainage discontinuation.
Time Frame: Date of chest tube drainage discontinuation, approximately 11 days after surgery
Population: Intention to Treat compared to colchicine per protocol
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Colchicine Intention to Treat: All patients entered the intended protocol where Colchicine was empirically given 0.6mg once daily to postoperative Fontan patients starting on postoperative day 2 and ending 1 day after chest tubes were removed or for a maximum of 4 weeks.
  This group were all of those who began the protocol, whether they completed it or not.
- Colchicine Per Protocol: All patients entered the intended protocol where Colchicine was empirically given 0.6mg once daily to postoperative Fontan patients starting on postoperative day 2 and ending 1 day after chest tubes were removed or for a maximum of 4 weeks.
  These patients completed the entire protocol.
Arm/Group | Colchicine Intention to Treat | Colchicine Per Protocol
Number analyzed (Participants) | 9 | 5
days | 7.5 [5.75 to 9] | 6 [4.5 to 7]

6. Secondary Outcome: Difference of Duration of Pleural Drainage of Two Groups, in Empiric Treatment With Colchicine Compared to a Cohort of Fontan Patients Not Treated With Colchicine
Description: Duration is measured in days, from date of Fontan surgery to chest tube drainage discontinuation
Time Frame: Date of chest tube drainage discontinuation, approximately 11 days after surgery
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Colchinine Intention to Treat: All patients entered the intended protocol where Colchicine was empirically given 0.6mg once daily to postoperative Fontan patients starting on postoperative day 2 and ending 1 day after chest tubes were removed or for a maximum of 4 weeks.
  These participants were in the trial at least initially, but not all completed the protocol.
Arm/Group | Colchicine Per Protocol | Colchinine Intention to Treat | Historical Controls
Number analyzed (Participants) | 5 | 9 | 25
days | 6 [4.5 to 7] | 7.5 [5.8 to 9] | 10 [7 to 11]
Statistical Analysis 1: Comparison: Colchicine Per Protocol vs Historical Controls; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Colchinine Intention to Treat vs Historical Controls; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Hospital Length of Stay as Measured in Postoperative Fontan Patients Treated Empirically With Colchicine
Description: Measured in days, from date of Fontan surgery to chest tube drainage discontinuation
Time Frame: Hospital discharge at study completion, approximately 2 weeks after surgery
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Colchicine Intention to Treat: All patients entered the intended protocol where Colchicine was empirically given 0.6mg once daily to postoperative Fontan patients starting on postoperative day 2 and ending 1 day after chest tubes were removed or for a maximum of 4 weeks.
  These patients were all those assigned to the protocol whether they completed it or not.
Arm/Group | Colchicine Intention to Treat | Colchicine Per Protocol
Number analyzed (Participants) | 9 | 5
days | 9 [6.5 to 11] | 7 [5.5 to 8.5]

8. Secondary Outcome: Difference in Hospital Length of Stay
Description: Measured in days compared to historical controls
Time Frame: Hospital discharge at study completion, approximately 2 weeks after surgery
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Colchicine Intention to Treat: All patients entered the intended protocol where Colchicine was empirically given 0.6mg once daily to postoperative Fontan patients starting on postoperative day 2 and ending 1 day after chest tubes were removed or for a maximum of 4 weeks.
  All of these participants began the protocol, but not all these participants completed the protocol.
Arm/Group | Colchicine Per Protocol | Colchicine Intention to Treat | Historical Controls
Number analyzed (Participants) | 5 | 9 | 25
days | 7 [5.5 to 8.5] | 9 [6.5 to 11] | 11 [9 to 13]
Statistical Analysis 1: Comparison: Colchicine Per Protocol vs Historical Controls; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Colchicine Intention to Treat vs Historical Controls; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: from initiation of study through 5-14 days after last dose of colchicine (generally 12 -21 days)
Description: As noted earlier under Participant Flow, historical controls were not considered enrolled in this trial. Further, the historical control information comes from an observational study in which Adverse Events were not collected. Thus, historical control data is not presented.
Arm/Group | Colchicine
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colchicine (N=9)
nausea (Gastrointestinal disorders) | 5
increase in creatinine (Renal and urinary disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
hepatic dysfunction (Hepatobiliary disorders) | 1
vomiting (Gastrointestinal disorders) | 5
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
loose stool (Gastrointestinal disorders) | 1
abdominal pain (Gastrointestinal disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT03575572/Prot_SAP_000.pdf